CLINICAL TRIAL: NCT07363109
Title: Prevention of Hypotension During Elective Cesarean Section Under Spinal Anaesthesia With Fixed-rate Metaraminol Infusion Versus Fixed-rate Norepinephrine Infusion: A Double-blind Randomised Controlled Clinical Trial.
Brief Title: Comparison of the Efficacy of Continuous Metaraminol Infusion Versus Continuous Norepinephrine Infusion for the Prevention of Hypotension During Cesarean Section Under Spinal Anaesthesia. A Randomised Controlled Trial.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aretaieion University Hospital (Other)
Responsible Party: Principal Investigator, Adamantia Gkaniou, Resident anaesthesiologist, MD, MSc, Aretaieion University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 719/28-11-2025
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Hypotension After Spinal Anesthesia; Hypotension During Cesarean Delivery
Keywords: metaraminol; norepinephrine; prevention of hypotension; cesarean section; maternal hemodynamics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metaraminol group (Active Comparator)
  Interventions: Procedure: Metaraminol infusion
- Norepinephrine group (Active Comparator)
  Interventions: Procedure: Norepinephrine infusion

INTERVENTIONS:
Procedure: Metaraminol infusion — In parturients allocated to the metaraminol group, a metaraminol infusion (30 mL/h corresponding to 100 μg/min) will be initiated as soon as spinal anaesthesia is established.
  Arms: Metaraminol group
Procedure: Norepinephrine infusion — In parturients allocated to the norepinephrine group, a norepinephrine infusion (30 mL/h corresponding to 4 μg/min) will be initiated as soon as spinal anaesthesia is established.
  Arms: Norepinephrine group

SUMMARY:
The aim of this double-blind randomised study will be to compare a fixed-rate prophylactic metaraminol infusion to a fixed-rate prophylactic norepinephrine infusion during elective cesarean section under combined spinal-epidural anaesthesia.

DETAILED DESCRIPTION:
Spinal anaesthesia is the anaesthetic technique of choice for elective cesarean section.

Spinal anaesthesia can be complicated by hypotension, with incidence exceeding 80% occasionally. Hypotension can lead to nausea, emesis and a subjective feeling of discomfort due to cerebral hypoperfusion. If left untreated, severe or sustained hypotension can lead to decreased uteroplacental flow and fetal distress of premature or compromised fetuses while severe complications to the parturient might ensue, such as loss of consciousness, aspiration, apnea or cardiac arrest.

Prophylactic vasoconstrictor infusion is an effective strategy for preventing maternal hypotension during regional anaesthesia. Phenylephrine is widely used because it acts quickly and causes less neonatal acidosis than ephedrine, but high doses may reduce maternal cardiac output. Norepinephrine and metaraminol, a sympathomimetic amine that acts both directly and indirectly, mainly by stimulating alpha-1-adrenergic receptors, with a weak effect on beta-receptors, have emerged as potential alternatives. While the optimal norepinephrine infusion dose has been defined in several studies, research on metaraminol remains limited, with insufficient data on its ideal dosing and efficacy in obstetrics. Most comparative studies evaluate metaraminol against phenylephrine-some suggesting better fetal acid-base outcomes-but no studies directly compare metaraminol with norepinephrine. Further research is therefore needed before metaraminol can be routinely recommended in obstetric anaesthesia.

This study will include pregnant adults who are normotensive, without complications, with a single pregnancy, who are not in active labor, and who are scheduled to undergo an elective cesarean section at the Gynecology-Obstetrics Clinic of Aretaieion Hospital.The study will use randomized, concealed allocation to assign participants to receive either metaraminol or norepinephrine infusions. Study group allocation will take place according to a computer-generated sequence of random numbers. A non-involved healthcare professional will reveal each participant's assignment, and a nurse will prepare identical 50 mL syringes labeled "study infusion," containing the drug at concentrations that deliver either 100 µg/min (200 µg/mL at 30 mL/h) of metaraminol or 4 µg/min (8 µg/mL at 30 mL/h) of norepinephrine. The anaesthesiologist, patient, and data analyst will remain blinded to group allocation.

All parturients will receive standard pre-anesthetic evaluation and standard hemodynamic monitoring will be applied. Next, on the hand opposite the one with the cuff for measuring NIBP, a special finger cuff connected to the Edwards Lifesciences ClearSight system will be placed on the index, middle, or ring finger. The ClearSight system from Edwards Lifesciences is a non-invasive medical system that allows continuous monitoring of blood pressure (cBP), as well as a range of other hemodynamic parameters such as cardiac output (CO), stroke volume (SV), and systemic vascular resistance (SVR).

Baseline systolic arterial pressure will be considered the average of three consecutive measurements that will not differ more than 10% among them.

All parturients will have a peripheral intravenous catheter placed in the upper extremity after baseline hemodynamic measurements are recorded. The peripheral venous catheter in the arm without the cuff will be connected via a three-way stopcock and a small-volume tube to an infusion syringe placed in an electronic infusion pump in standby mode. The syringe will contain the corresponding vasoactive drug "study infusion." At the same time, infusion of Ringer/Lactate solution at a dose of 3 mL/kg/h will begin through the study infusion line (pre-loading) before the regional procedure.

A standard spinal anaesthetic consisting of ropivacaine 0.75% 1.8 mL plus fentanyl 10 μg will be administered in the left lateraL position at the L3-4 or L4-5 vertebral interspace. The study infusion medication (either metaraminol or norepinephrine, depending on group allocation) will be started at the same time cerebrospinal fluid is obtained, immediately before injection of spinal medications. After the intrathecal injection, patients will placed in the supine position with a left lateral tilt to provide left uterine displacement and to prevent aortocaval compression. The spinal sensory level will be tested bilaterally to ensure a T4 dermatomal level before surgical incision.

Hemodynamic parameters [systolic blood pressure (SAP), diastolic blood pressure (DAP), mean arterial pressure (MAP), heart rate (HR), cardiac output (CO), stroke volume (SV), and systemic vascular resistance (SVR)] will be recorded by a specially trained, experienced anaesthesiologist at specific time points during the procedure: baseline (T0), initiation of the study drug infusion (T1), placement in the supine position after subarachnoid administration (T2), sympathetic blockade at the T4 level (T3), start of surgery (T4), delivery of the newborn (T5), 5 minutes after administration of the oxytocin bolus (T6), end of surgery (T7).

Requirements for additional vasoactive agents and any adverse effects and complications in the mother's health will also be recorded.

Hypotension will be defined as SAP < 80% of baseline, hypertension as SAP > 120% of baseline, and bradycardia as HR < 60 bpm. In case of hypotension combined with HR > 80/min, a dose of 50 μg of phenylephrine will be administered, while when hypotension is combined with HR < 80/min, a dose of 5 mg of ephedrine will be administered. Episodes of hypertension (SAP > 120% of baseline) will be treated by reducing the infusion of the "study drug" by half (15 ml/h) while if blood pressure rises to levels >130% of the baseline value, administration of the vasoconstrictor solution will be discontinued. In case of bradycardia (HR < 60 bpm) in combination with SAP within 80%-120% of baseline or hypertension, the infusion of the "study drug" will be discontinued without the administration of atropine. When HR < 55 bpm in combination with hypotension (SAP value < 80% of baseline) or in case of HR < 50 bpm regardless of the degree of hypotension, 0.6 mg of atropine will be administered.

Neonatal pH values in the first blood gas sample immediately after birth will be recorded, as well as the Apgar score at 1 and 5 minutes after birth.

The clinical interest of the study lies in determining whether the use of metaraminol is superior to the administration of norepinephrine as a vasoconstrictor during cesarean section and to what extent it ensures hemodynamic stability of the mother and a more favorable metabolic profile of the newborn.

ELIGIBILITY:
Inclusion Criteria:

adult parturients, singleton gestation, elective cesarean section

Exclusion Criteria:

ASA >II, age <18 years, Body Mass Index (BMI) >40 kg/m2, body weight <50 kg, body weight>100 kg, height<150 cm, height>180 cm, multiple gestation, fetal abnormality, fetal distress, active labor, emergency CT, cardiovascular disease or cerebrovascular disease, pre-existing or pregnancy-induced hypertension, use of antihypertensive medication during pregnancy, preeclampsia, any contraindication for regional anesthesia, such as thrombocytopenia or coagulation disorder, communication or language barriers, lack of informed consent

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-02 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
incidence of hypotension | intraoperative
  any occurrence of hypotension throughout the operation will be recorded (SAP < 80% of baseline)
number of hypotensive episodes in the pregnant woman | intraoperativre
  the number of hypotensive episodes (SAP < 80% of baseline)throughout the operation will be recorded
incidence of bradycardia | intraoperative
  any incidence of HR < 60/min will be recorded

SECONDARY OUTCOMES:
need for vasoconstrictor | intraoperative
  parturient needed or not vasoconstrictor during the operation
type of bolus vasopressor administered | intraoperative
  phenylephrine verus ephedrine
number of bolus doses of vasoconstrictor administered | intraoperative
  number of provided interventions to maintain systolic blood pressure within the set limits will be recorded
total dose of vasoconstrictor administered | intraoperative
  total dose in mg for ephedrine or μg for phenylephrine
need for administration of atropine | intraoperative
  parturient needed or not atropine during the operation
incidence of hypertension | intraoperative
  any incidence of systolic blood pressure >120% of baseline will be recorded
need for differentiation in the basic infusion rate of the vasopressor solution | intraoperative
  due to the occurrence of bradycardia or reactive hypertension
incidence of nausea/vomiting | intraoperative
  incidence of nausea and vomiting throughout the operation
Incidence of dizziness, discomfort, and shivering | intraoperative
  Incidence of dizziness, discomfort, and shivering through the operation
neonatal Apgar score | 1 min and 5 min post delivery
  Neonatal Apgar score will be recorded at 1 min and at 5 min after delivery. The Apgar score is determined by evaluating the newborn baby on five simple criteria on a scale from zero to two, then summing up the five values thus obtained. The resulting Apgar score ranges from zero to 10. Scores 7 and above are generally normal; 4 to 6, fairly low; and 3 and below are generally regarded as critically low and cause for immediate resuscitative efforts.
neonatal blood gases | 1 min post delivery
  fetal cord blood analysis will be performed immediately post-delivery
glucose in neonatal blood | 1 min post delivery
  glucose will be measured in the cord blood gas sample taken immediately post-delivery

CONTACTS AND LOCATIONS:
Overall Officials: Kassiani Theodoraki, Study Director — Aretaieion University Hospital, National and Kapodistrian University of Athens

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McDonnell NJ, Paech MJ, Muchatuta NA, Hillyard S, Nathan EA. A randomised double-blind trial of phenylephrine and metaraminol infusions for prevention of hypotension during spinal and combined spinal-epidural anaesthesia for elective caesarean section. Anaesthesia. 2017 May;72(5):609-617. doi: 10.1111/anae.13836. Epub 2017 Mar 3. PMID 28255987
- [Background] Chao E, Sun HL, Huang SW, Liao JH, Ma PL, Chen HC. Metaraminol use during spinal anaesthesia for caesarean section: a meta-analysis of randomised controlled trials. Int J Obstet Anesth. 2019 Aug;39:42-50. doi: 10.1016/j.ijoa.2019.01.009. Epub 2019 Jan 25. PMID 30772119
- [Background] Lyu W, Zhang Z, Li C, Wei P, Feng H, Zhou H, Zheng Q, Zhou J, Li J. Intravenous initial bolus during prophylactic norepinephrine infusion to prevent spinal hypotension for cesarean delivery: A randomized controlled, dose-finding trial. J Clin Anesth. 2024 Oct;97:111562. doi: 10.1016/j.jclinane.2024.111562. Epub 2024 Jul 23. PMID 39047530
- [Background] Xiao F, Xu WP, Yao HQ, Fan JM, Chen XZ. A Randomized Double-Blinded Dose-dependent Study of Metaraminol for Preventing Spinal-Induced Hypotension in Caesarean Delivery. Front Pharmacol. 2021 May 12;12:608198. doi: 10.3389/fphar.2021.608198. eCollection 2021. PMID 34054513
- [Background] Ngan Kee WD, Khaw KS, Ng FF. Comparison of phenylephrine infusion regimens for maintaining maternal blood pressure during spinal anaesthesia for Caesarean section. Br J Anaesth. 2004 Apr;92(4):469-74. doi: 10.1093/bja/aeh088. Epub 2004 Feb 20. PMID 14977792
- [Background] Ngan Kee WD. Prevention of maternal hypotension after regional anaesthesia for caesarean section. Curr Opin Anaesthesiol. 2010 Jun;23(3):304-9. doi: 10.1097/ACO.0b013e328337ffc6. PMID 20173633
- [Background] Fitzgerald JP, Fedoruk KA, Jadin SM, Carvalho B, Halpern SH. Prevention of hypotension after spinal anaesthesia for caesarean section: a systematic review and network meta-analysis of randomised controlled trials. Anaesthesia. 2020 Jan;75(1):109-121. doi: 10.1111/anae.14841. Epub 2019 Sep 18. PMID 31531852
- [Background] Bower JR, Kinsella SM. Preventing and treating hypotension during spinal anaesthesia for caesarean section. BJA Educ. 2020 Nov;20(11):360-361. doi: 10.1016/j.bjae.2020.08.001. Epub 2020 Sep 9. No abstract available. PMID 33456918
- [Background] Gizzo S, Di Gangi S, Noventa M, Bacile V, Zambon A, Nardelli GB. Women's choice of positions during labour: return to the past or a modern way to give birth? A cohort study in Italy. Biomed Res Int. 2014;2014:638093. doi: 10.1155/2014/638093. Epub 2014 May 15. PMID 24955365
- [Background] Nguyen-Lu N, Carvalho JC, Kingdom J, Windrim R, Allen L, Balki M. Mode of anesthesia and clinical outcomes of patients undergoing Cesarean delivery for invasive placentation: a retrospective cohort study of 50 consecutive cases. Can J Anaesth. 2016 Nov;63(11):1233-44. doi: 10.1007/s12630-016-0695-x. Epub 2016 Jul 21. PMID 27443374
- [Background] Kim WH, Hur M, Park SK, Yoo S, Lim T, Yoon HK, Kim JT, Bahk JH. Comparison between general, spinal, epidural, and combined spinal-epidural anesthesia for cesarean delivery: a network meta-analysis. Int J Obstet Anesth. 2019 Feb;37:5-15. doi: 10.1016/j.ijoa.2018.09.012. Epub 2018 Sep 27. PMID 30415797
- [Background] Theodoraki K, Hadzilia S, Valsamidis D, Stamatakis E. Prevention of hypotension during elective cesarean section with a fixed-rate norepinephrine infusion versus a fixed-rate phenylephrine infusion. Alpha double-blinded randomized controlled trial. Int J Surg. 2020 Dec;84:41-49. doi: 10.1016/j.ijsu.2020.10.006. Epub 2020 Oct 17. PMID 33080415
- [Background] Sumikura H, Niwa H, Sato M, Nakamoto T, Asai T, Hagihira S. Rethinking general anesthesia for cesarean section. J Anesth. 2016 Apr;30(2):268-73. doi: 10.1007/s00540-015-2099-4. Epub 2015 Nov 19. PMID 26585767
- [Background] Iddrisu, M., Khan, Z.H. Anesthesia for cesarean delivery: general or regional anesthesia-a systematic review. Ain-Shams J Anesthesiol 13, 1 (2021). https://doi.org/10.1186/s42077-020-00121-7
- [Background] Angolile CM, Max BL, Mushemba J, Mashauri HL. Global increased cesarean section rates and public health implications: A call to action. Health Sci Rep. 2023 May 18;6(5):e1274. doi: 10.1002/hsr2.1274. eCollection 2023 May. PMID 37216058
- [Background] Ghaffari S, Dehghanpisheh L, Tavakkoli F, Mahmoudi H. The Effect of Spinal versus General Anesthesia on Quality of Life in Women Undergoing Cesarean Delivery on Maternal Request. Cureus. 2018 Dec 11;10(12):e3715. doi: 10.7759/cureus.3715. PMID 30788204